CLINICAL TRIAL: NCT01710852
Title: A Phase 2 Study to Assess the Antiarrhythmic and Symptomatic Effect of the Second Generation Antisense Oligonucleotide ISIS 329993 Targeting CRP in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Antiarrhythmic and Symptomatic Effect of ISIS CRP Rx Targeting CRP in Paroxysmal Atrial Fibrillation
Acronym: ASET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 329993-CS6
Record Dates: First submitted 2012-10-09; First posted 2012-10-19 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; AF
MeSH Terms: conditions — Atrial Fibrillation | interventions — ISIS 329993

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): ISIS CRP Rx followed by Placebo
  Interventions: Drug: ISIS CRP Rx; Drug: Placebo
- Group B (Experimental): Placebo followed by ISIS CRP Rx
  Interventions: Drug: ISIS CRP Rx; Drug: Placebo

INTERVENTIONS:
Drug: ISIS CRP Rx
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate whether treatment with ISIS CRP Rx can reduce AF (Atrial Fibrillation) burden (percentage of time spent in AF) in subjects with paroxysmal AF

ELIGIBILITY:
Inclusion Criteria:

* Male of female; age over 18 years
* Dual chamber permanent pacemaker implanted
* Confirmed diagnosis of paroxysmal atrial fibrillation with an AF burden of 1 to 50%, as derived from pacemaker diagnostic algorithms
* Able to have pacemaker antiarrhythmic algorithms turned off for the duration of the study
* Able to discontinue all Class I and III antiarrhythmic medication for the duration of the study
* Therapeutically anticoagulated with warfarin or dabigatran, and anticipated to be for duration of the study
* High sensitivity C-Reactive Protein (hsCRP) between 2 and 10 mg/L (inclusive)

Exclusion Criteria:

* Clinically significant abnormalities in medical history, physical examination, or screening laboratory results that would render a subject unsuitable for inclusion
* NYHA class III/IV heart failure
* Impaired left ventricular function of less than 45% determined by echocardiography within 3 months of screening
* Moderate or greater mitral regurgitation assessed by echocardiography within 3 months of screening
* Permanent AF
* Continuous Amiodarone therapy within 90 days prior to Study Day 1
* Treatment with another Study Drug, biological agent, or device within one-month of screening, or five half-lives of study agent, whichever is longer
* Use of systemic corticosteroids or other anti-inflammatory medications including non-steroidal anti-inflammatory drugs (NSAIDs)
* Use of statins, ACE inhibitors or AT-receptor antagonists unless on a stable regimen for at least 3 months prior to dosing and will remain on a stable regimen for the duration of the study
* Uncontrolled hypertension (BP >160/100)
* Current or expected use of any anticoagulant apart from warfarin or dabigatran

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
AF burden reduction | 113 Days
  Burden measured as percentage of time spent in AF as derived from continuous pacemaker monitoring

SECONDARY OUTCOMES:
To assess the effect of ISIS CRP Rx on the: | 113 Days
  * total number of AF episodes
  * average duration of AF per episode
  * average sinus rhythm duration
  * atrial and ventricular rate during AF episodes
To assess the effect of ISIS CRP Rx on ventricular rate during sinus rhythm | 113 Days
To assess the effect of ISIS CRP Rx on measures of Quality of Life | 113 Days
To assess whether treatment with ISIS CRP Rx reduces hsCRP in subjects with paroxysmal AF | 113 Days
  Change from Baseline will be compared for each treatment period
To assess the safety of ISIS CRP Rx in subjects with paroxysmal AF | 113 Days
  Incidence rates of all Adverse Events will be tabulated by MedRA system Organ Class and by MedRA Term for each treatment group. Lab Tests, Vital Signs, And ECG Parameters will be summarized by study visit for each treatment group.
To assess the tolerability of ISIS CRP Rx in subjects with paroxysmal AF | 113 Days
  Incidence rates of all Adverse Events will be tabulated by MedRA system Organ Class and by MedRA Term for each treatment group. Lab Tests, Vital Signs, And ECG Parameters will be summarized by study visit for each treatment group.
To assess the pharmacokinetics of ISIS CRP Rx in subjects with paroxysmal AF | 113 Days
  Trough levels of ISIS CRP Rx will be assessed at intervals throughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- Eastbourne General Hospital - Cardiology Department, Eastbourne, East Sussex, United Kingdom